CLINICAL TRIAL: NCT04165668
Title: Wellbeing and Stress Among Lay Responders Dispatched to Suspected Out-of-hospital Cardiac Arrests
Brief Title: Wellbeing and Stress Among Mobile Phone Dispatched Lay Responders
Status: Terminated | Type: Observational
Why Stopped: Due to the COVID-19 Pandemic.
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Vastra Gotaland Region (Other Government); Uppsala University (Other); ESCAPE-NET investigators (Unknown)
Responsible Party: Principal Investigator, Mattias Ringh, Principal Investigator, Karolinska Institutet
Other Study IDs: Karolinskal007
Record Dates: First submitted 2019-11-11; First posted 2019-11-18 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Stress, Psychological; Post-traumatic Stress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dispatched lay responders: Nearby mobile phone located and dispatched lay responders who reached the place of the suspected OHCA before EMS and first responders (fire and police services).
  Interventions: Other: Exposure: First on scene
- Non-dispatched lay responders: Nearby mobile phone located lay responders who have neither actively, nor technically responded due to either human or technical factors.

INTERVENTIONS:
Other: Exposure: First on scene — To be first on scene for resuscitation at the suspected out-of hospital cardiac arrest, before EMS and first responders (fire and police services)
  Groups: Dispatched lay responders

SUMMARY:
The aim of this study is to provide detailed information on state of mind, psychological wellbeing and stress for lay responders dispatched to suspected OHCA via a mobile phone application.

The Heartunner system is a mobile phone positioning system for dispatch of CPR-trained lay volunteers to nearby suspected out-of-hospital cardiac arrests (OHCAs). After downloading of a mobile phone application (The Heartrunner application), and given consent of participation, the lay responders are dispatched to nearby suspected OHCA. The lay responders are either dispatched directly to the scene of the suspected OHCA to perform CPR, or to fetch the nearest AED. The location of the OHCA and available AEDs are displayed on a map, facilitated by the Heartrunner application. The Heartrunner system is studied through "The SAMBA-trial" on clinical outcomes for OHCA patients (ClinicalTrials.gov Identifier: NCT02992873).

The psychological effects among the lay responders will be evaluated with an online survey adjacent to dispatch and after 4-6 weeks. The results of the survey will be compared both intra-individual, and to a control group of not dispatched lay responders within the Heartrunner system. Descriptive statistics regarding interventions, age, gender and former experience will also be presented.

DETAILED DESCRIPTION:
Please see the attacehd study protocol for details

ELIGIBILITY:
Inclusion Criteria:

* Mobile phone dispatched lay responders who reached the scene a suspected cardiac arrest.
* Located lay responders who was not dispatched due to technical or human reasons (no feedback from app to system).

Exclusion Criteria:

* Mobile Phone Lay responders who declined the mission for dispatch to a suspected cardiac arrest.
* Mobile Phone Lay responders that already answered the survey.
* Mobile phone dispatched lay responders who accepted the mission but was aborted due to distance or did not reach the scene.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lay responders participating as volunteers in the Heartrunner system in regions of Stockholm and Västra Götaland.
Sampling Method: Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Change in Level of stress at 4 weeks | At 90 minutes and 4 at weeks
  Swedish Core Affect Scale (SCAS);The measure of state of mind will be done on 12 affective scales of adjective pairs that range from 1-9. For example: anxious (1) to calm (9), pessimistic (1) to optimistic (9) etc. High numbers on adjectives indicating activation, as well as measures on "Anxious", "tense" and "nervous" will be regarded as (negative) stress whereas "Interested" "engaged" and "optimistic" will be regarded as (positive) stress.

SECONDARY OUTCOMES:
Level of post traumatic stress symptoms | At 90 minutes and 4 at weeks
  PCL checklist, short form with 6 items each ranging from 1 to 5. Max is 30 points and a positive screen is a score of ≥ 14 points.
Level of wellbeing | At 4 weeks
  WHO index, 5 questions each ranging from 5-1 with a maximum of 100 points were higher values indicate good wellbeing. A score below 14 indicates poor wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Ringh, MD PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Västra Götaland, Gothenburg
  - Stockholm, Sweden, Stockholm